CLINICAL TRIAL: NCT06578871
Title: Surgery for the Unknown Primary in the Era of p16-positive Oropharyngeal Squamous Cell Carcinoma: Reducing Ionizing Radiation (SUPERIOR): A Randomized Trial
Brief Title: Surgery and Reducing Ionizing Radiation of the Unknown Primary
Acronym: SUPERIOR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Dr. Jake Jervis-Bardy (Unknown); Dr. David Palma (Unknown); Dr. Adam Mutsaers (Unknown)
Responsible Party: Principal Investigator, Adrian Mendez, Study Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15080; 5007 (Other: OCREB)
Record Dates: First submitted 2024-08-14; First posted 2024-08-29 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma; HPV Positive Oropharyngeal Squamous Cell Carcinoma
Keywords: HPV-Mediated PUK; Head and Neck Cancer; P16+; Radiation Therapy; Oropharyngeal Cancer; Squamous Cell Carcinoma; Transoral Robotic Surgery (TORS); Mucosal Radiation; SUPERIOR Trial
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Oropharyngeal Neoplasms; Carcinoma, Squamous Cell | interventions — Radiotherapy, Intensity-Modulated; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: This is a randomized phase II study. Patients will be randomized between current standard of care treatment (Arm 1) vs. omission of radiation mucosal surfaces (Arm 2) in a 1:2 ratio.
Who Masked: Outcomes Assessor
Masking Description: The SUPERIOR trial employs a 1:2 randomization ratio using a permuted block design with block sizes known only to the statistician. Stratification factors include smoking status (>10 pack-years vs. ≤10 pack-years) and pathologic nodal burden (1 node positive vs. >1 node positive). Although participants and treating clinicians are aware of the treatment allocations, outcome assessors and data analysts are blinded to the treatment arms to ensure unbiased assessment and analysis of trial results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1: Standard of Care Treatment (Active Comparator): Radiotherapy to Ipsilateral Neck and to risk Mucosa
  There are two possible dose levels:
  * 60 Gy in 30 fractions over 6 weeks (CTV60)
    o This applies to the dissected levels of the neck
  * 54 Gy in 30 fractions over 6 weeks (CTV54)
    * This applies to the mucosal surfaces. Patients randomized to Arm 2 will not have the mucosal surfaces treated
  Interventions: Radiation: Intensity Modulated Radiotherapy (IMRT) to Mucosa at Risk; Procedure: Surgical Intervention; Radiation: Intensity Modulated Radiotherapy (IMRT) to Ipsilateral Neck
- Arm 2: Omission of IMRT to Risk Mucosa but conditional IMRT to Neck (Experimental): * If N1 with single node <= 3cm, no further treatment
  * If multiple ipsilateral nodes or single ipsilateral node >3 cm, radiation to Neck only
  Interventions: Procedure: Surgical Intervention; Radiation: Intensity Modulated Radiotherapy (IMRT) to Ipsilateral Neck

INTERVENTIONS:
Radiation: Intensity Modulated Radiotherapy (IMRT) to Mucosa at Risk — Patients in Arm 1, after the surgical procedure, will receive radiotherapy to the at-risk mucosa.
  Arms: Arm1: Standard of Care Treatment
Procedure: Surgical Intervention — These patients will undergo Neck dissection, TORS tonsillectomy (unilateral vs bilateral tonsillectomy at the discretion of the treating physician) + ipsilateral tongue base mucosectomy.
Radiation: Intensity Modulated Radiotherapy (IMRT) to Ipsilateral Neck — For Arm1, after the surgical procedure, the patients will receive radiotherapy to the ipsilateral neck. For Arm2, the patients will only receive IMRT to neck, if multiple ipsilateral nodes or single ipsilateral node >3 cm is observed

SUMMARY:
About 3% of people with head and neck cancer have cancer in their lymph nodes, but doctors are unable to find the primary tumour. This situation has become more common due to human papillomavirus (HPV), a virus linked to certain cancers. Generally, patients with HPV-related cancers have a good outlook, with around 90% surviving for at least five years.

Recent advancements in medical technology, such as advanced imaging and specialized surgeries, have significantly improved doctors' ability to find these hidden tumours. These techniques can locate the primary tumour in 70-80% of cases. If the tumour remains undetected, it could be very small or potentially eliminated by the body's immune system.

The best way to treat this type of cancer is still debated. Current treatment options include surgery to remove lymph nodes or radiation therapy. There is no clear agreement on which areas should receive radiation. Often, surgery is performed on one side of the throat to try and locate the tumour's origin.

Researchers are exploring ways to minimize the harmful side effects of treatment. Some studies suggest that surgery alone might be sufficient for patients with small tumours in their neck, but more research is needed. Another important question is whether radiation needs to cover the entire throat area. Recent findings suggest that omitting radiation from some areas might reduce side effects such as difficulty swallowing and dry mouth.

The SUPERIOR trial aims to investigate whether reducing the amount of radiation can still be effective and improve patients' quality of life. The study also examines whether surgery alone is adequate for certain patients with HPV-related cancers.

DETAILED DESCRIPTION:
Approximately 3% of all head and neck squamous cell carcinoma (SCC) patients present with nodal disease from an unknown primary (PUK). The incidence of PUK has increased in tandem with the rise of human papillomavirus (HPV)-mediated oropharyngeal SCC (OPSCC). HPV-mediated PUK now represents at least half of the head and neck PUK population, with an excellent prognosis and approximately 90% 5-year overall survival (OS).

The work-up for PUK has significantly improved with the introduction of positron emission tomography (PET) imaging and transoral robotic surgery (TORS). PET identifies at least 40% of primaries in PUK patients when clinical and radiological work-up is negative, and TORS has a higher primary identification rate (70%-80%). Current guidelines recommend tonsillectomy and tongue base mucosectomy in the work-up of PUK patients.

Definitive management of HPV-mediated PUK remains controversial, with curative options including primary neck dissection ± adjuvant therapy or primary radiotherapy ± concurrent chemotherapy. Treatment morbidity is significant, despite the excellent outcomes (90% 5-year OS). Key issues include the choice of initial treatment modality and whether to treat mucosal surfaces with radiation prophylactically.

Current guidelines recommend single-modality surgery (neck dissection) for low-volume neck disease. This recommendation is based on studies suggesting low primary emergence rates (1.5%-7%) and outcomes comparable to non-surgical treatment paradigms. Evidence from early-stage OPSCC supports surgery alone as a safe option for HPV-mediated PUK.

A critical question is whether to irradiate mucosal surfaces when using radiotherapy for HPV-mediated PUK. Emerging data suggest that omitting mucosal radiation has a very low risk (<5%) of primary tumour emergence, potentially improving long-term quality of life and reducing toxicities like dysphagia and xerostomia. Several retrospective studies support the safety and reduced toxicity of involved neck radiotherapy without mucosal irradiation.

This trial is specifically designed with an upfront neck dissection alongside tonsillectomy and tongue base mucosectomy. Combining an upfront therapeutic neck dissection with the final stage of the diagnostic work-up has several benefits. Surgically treating the neck in selected patients during tonsillectomy and tongue base mucosectomy accelerates treatment, avoids additional delays, reduces costs to healthcare institutions, and prevents the need for a second surgery if no primary is identified. The addition of neck dissection to tonsillectomy and tongue base mucosectomy also involves relatively minor additional surgical morbidity in the context of a patient already undergoing pharyngeal surgery. In some instances, upfront surgical treatment of the neck may complete definitive treatment at the earliest opportunity. Patients with intermediate-volume neck disease, who require dual-modality treatment, also benefit from no further surgical delay and can proceed to radiotherapy following a single surgical encounter. An upfront neck dissection is also the gold standard for lymph node evaluation and may down-stage patients into a unimodality approach, thereby avoiding additional toxicity. For example, if imaging suggests multiple involved ipsilateral nodes in an HPV-mediated PUK patient, conventional treatment would involve dual-modality therapy. Pathological staging may down-stage this patient into a unimodality paradigm, sparing them significant toxicity.

In this randomized phase II trial, the study team hypothesizes that omitting mucosal radiation will lead to improved quality of life, decreased toxicity, and low rates of primary tumour emergence. Further, the researchers hypothesize that neck dissection alone for low-volume HPV-mediated PUK will result in excellent oncologic and functional outcomes.

The main objective is to assess the impact of omitting mucosal radiation on oncologic outcomes, toxicity, functional outcomes, and quality of life (QOL) in patients with p16-positive PUK.

The primary endpoint is to determine the rate of primary emergence of a mucosal p16-positive SCC in the upper aerodigestive tract compared to historical controls.

The secondary endpoints include:

Quality of life (using MDADI, EORTC QLQ-C30 and H&N35, EQ-5D-5L, NDII) Overall survival (OS) Disease-free survival Regional recurrence within the neck Distant recurrence outside the upper aerodigestive tract and neck levels Rate of salvage treatment for primary emergence Rate of unsalvageable primary emergence Rate of percutaneous feeding tube insertion and use at 1 year Swallowing function (DIGEST score, FOIS) Toxicity (CTCAE version 5) Patients will be randomized 1:2 between the standard of care (Arm 1) and omission of radiation to mucosal surfaces (Arm 2).

Combining neck dissection with tonsillectomy and tongue base mucosectomy accelerates treatment, reduces costs, and avoids additional surgery. This approach involves minor additional surgical morbidity and can complete definitive treatment at the earliest opportunity. Upfront neck dissection also allows for accurate lymph node evaluation and potential down-staging, thereby sparing patients from additional toxicity.

The SUPERIOR trial aims to determine whether omitting mucosal radiation improves quality of life and reduces toxicity in HPV-mediated PUK patients, while evaluating the efficacy of neck dissection alone for low-volume disease. The study seeks to establish evidence-based guidelines for the optimal management of HPV-mediated PUK.

ELIGIBILITY:
Inclusion criteria for the Registration phase

* p16 positive PUK SCC of the neck
* Age 18 years or older
* Willing to provide informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Clinical nodal stage N1, AJCC 8th edition (i.e. clinical unilateral nodal disease, none larger than 6 cm)
* Complete clinical work-up, including CT neck, physical examination with nasopharyngoscopy, and PET/CT, with no evidence of a primary tumor. The PET/CT scan must be without focal metabolic activity concerning for a primary tumor, in the opinion of the nuclear medicine physician. Metabolic activity, particularly in the tonsils and base of the tongue which is within normal physiologic range, does not exclude participation.

Inclusion criteria for the Randomization phase

* Completed ipsilateral tonsillectomy and base of tongue mucosectomy with no evidence of a primary tumor

  o Note, patients who had a PET/CT that was initially positive, and therefore not meeting criteria in 4.10, but panendoscopy with biopsies of the fluorodeoxyglucose (FDG)-avid areas do not show malignancy, can then be enrolled and would be returned the OR for a neck dissection prior to randomization
* Ipsilateral nodal disease on pathology with no evidence of extranodal extension

Exclusion Criteria:

* Radiological or pathological extra-nodal extension
* Epstein-Barr Virus (EBV)-positive
* Clinical nodal stage (i.e. before neck dissection) N2-3, AJCC 8th edition (ie. bilateral nodes or node >6cm)
* Pathological nodal stage (i.e. after neck dissection) pN3
* Prior history of head and neck cancer within 2 years
* Any other active invasive malignancy, except non-melanotic skin cancers, low-risk prostate cancer, and stage I-IVA papillary or follicular thyroid cancer
* Known metastatic disease
* Unable to complete QOL questionnaires
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint: Rate of Primary Emergence of Mucosal p16-Positive Squamous Cell Carcinoma | 2 years
  The primary endpoint of this clinical trial is to assess the rate at which a primary mucosal p16-positive squamous cell carcinoma (SCC) emerges in the upper aerodigestive tract (which includes the oral cavity, pharynx, or larynx) in patients with p16-positive PUK of the head and neck. This rate will be compared to a historical control to determine the impact of omitting mucosal radiation in these patients. The primary objective is to evaluate the oncologic outcomes associated with this treatment approach.

SECONDARY OUTCOMES:
MD Anderson Dysphagia Inventory (MDADI) | Assessed at baseline, 6 months, and 1 year post randomization
  MD Anderson Dysphagia Inventory (MDADI): Measures the impact of swallowing difficulties on a patient's daily life and emotional well-being.
  Scale Range: 20 to 100. Interpretation: Higher scores indicate a better outcome, reflecting better swallowing function and less impact on quality of life.
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Time Frame: Assessed at baseline, 6 months, and 1 year post randomization.
  Outcome Measure: General health status and overall quality of life in cancer patients, including physical functioning, role functioning, emotional functioning, and overall health.
  Scale Range: 0 to 100.
  Interpretation: Higher scores on functional scales and global health status indicate a better outcome. Higher scores on symptom scales indicate a worse outcome.
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck 35 (EORTC QLQ-H&N35) | Assessed at baseline, 6 months, and 1 year post randomization
  Outcome Measure: Head and neck cancer-specific symptoms and issues, particularly related to treatment effects.
  Scale Range: 0 to 100. Interpretation: Higher scores on symptom scales indicate a worse outcome, reflecting more severe symptoms or problems related to head and neck cancer.
European Quality of life (Euro-QoL) 5-Dimension 5-Level (EQ-5D-5L): Visual Analog Scale | Assessed at baseline, 6 months, and 1 year post randomization
  Outcome Measure: Health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  Scale Range: -0.281 to 1 (Index value) and 0 to 100 (Visual Analog Scale).
  Interpretation: For the Index value, higher scores indicate a better outcome (better health-related quality of life). For the Visual Analog Scale, higher scores indicate better perceived overall health.
Neck Dissection Impairment Index (NDII): | Assessed at baseline, 6 months, and 1 year post randomization
  Outcome Measure: Specific impairments related to neck dissection, including physical and functional issues in the neck area.
  Scale Range: 0 to 100.
  Interpretation: Higher scores indicate a better outcome, reflecting fewer impairments and better neck function.
Overall Survival | From the date of randomization until the date of death from any cause, assessed for a minimum of five years.
  Overall Survival (OS): Defined as the time from randomization until death or the last follow-up, whichever occurs first.
Disease Free Survival | From the date of randomization until the date of first documented disease recurrence or progression, or death from any cause, whichever occurs first, assessed for a minimum of five years.
  The time from randomization until the first occurrence of disease recurrence, death, or the last follow-up, whichever comes first.
Regional Recurrence | From the date of randomization until the date of first documented regional recurrence or until date of death from any cause, assessed throughout the study with a minimum follow-up of five years.
  The occurrence of recurrent cancer specifically within the nodal levels of the neck (levels I-VI).
Distant Recurrence | From the date of randomization until the date of first documented distant recurrence or until date of death from any cause, assessed throughout the study with a minimum follow-up of five years.
  The development of recurrent cancer outside the upper aerodigestive tract and neck levels.
Rate of Salvage Treatment for Primary Emergence | Assessed throughout the study, with follow-up for at least 5 years from randomization.
  The frequency of additional treatments (surgery ± radiotherapy) required for the emergence of a p16-positive primary mucosal tumour, with the intent of cure.
Rate of Unsalvageable Primary Emergence | From the date of randomization until the initiation of salvage treatment for primary emergence, assessed throughout the study with a minimum follow-up of five years.
  The frequency of emergence of a p16-positive primary mucosal tumour that cannot be treated with surgery or radiotherapy with the intent of cure.
Rate of Percutaneous Feeding Tube Insertion and Use | From the date of randomization through one year, with follow-up assessments at one year. Percutaneous feeding tube insertion and use will be recorded throughout this period.
  The frequency of percutaneous feeding tube insertion and the rate of feeding tube use 1 year after randomization.
Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) score | From the date of randomization, with swallowing function assessed at one year post-randomization.
  Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) score: Measures the severity of swallowing dysfunction particularly related to the impact of cancer treatment on swallowing ability. It evaluates changes in swallowing function as seen through imaging techniques, such as fluoroscopy or videofluoroscopy.
  Scale Used: Typically, the DIGEST score is a categorical scale with grades ranging from 0 to 4.
  Lower Scores: Indicate less severe swallowing dysfunction or no dysfunction. Higher Scores: Indicate more severe swallowing dysfunction, with a greater impact on the ability to eat and drink.
Functional Oral Intake Score (FOIS) | From the date of randomization, with swallowing function assessed at one year post-randomization.
  Functional Oral Intake Score (FOIS): Assesses the ability to consume food and liquids by mouth. It assesses how much and what type of food and liquids a patient can safely consume.
  Scale Used: The FOIS is a categorical scale with grades ranging from 1 to 7.
  Lower Scores: Indicate greater dependence on non-oral feeding methods or more restricted oral intake.
  Higher Scores: Indicate greater ability to consume a wide variety of foods and liquids by mouth, with fewer restrictions.
Toxicity : Assessment of Treatment-Related Adverse Events Using CTCAE v5.0 | Toxicity will be monitored throughout the study, with evaluations at regular intervals up to 1 year or until date of death, whichever comes first, post-randomization.
  Toxicity will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, which categorizes the severity and type of adverse effects experienced by patients.
  The assessment focuses on:
  Severity of Adverse Events: Evaluate the intensity of side effects related to treatment, ranging from mild to severe.
  Type of Adverse Events: Identifies specific side effects, such as nausea, fatigue, pain, and other treatment-related symptoms.
  Frequency and Duration: Monitors how often and for how long patients experience these adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian I Mendez, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's; Jake Jervis-Bardy, MD, Principal Investigator — Royal Adelaide Hospital
Locations (3):
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Adelaide, South Australia
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
In line with our commitment to transparency and scientific progress, we will share our study protocol, statistical analysis plan, and participant consent forms with the broader research community after receiving Research Ethics Board (REB) approval.
  Study Protocol: Details the trial's objectives, design, methodology, and operational aspects, including participant criteria, interventions, and outcomes.
  Statistical Analysis Plan: Outlines the methods and statistical techniques for analyzing trial data.
  Participant Consent Forms: Follow OCREB guidelines, detailing study risks, benefits, and participants' rights, ensuring transparency in the consent process.
  These documents will be available on ClinicalTrials.gov. Researchers can request access by contacting Dr. Adrian Mendez at adrian.mendez@lhsc.on.ca or Halema Khan at halema.khan@lhsc.on.ca.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available once we receive OCREB approval. Hopefully by November of 2024.
Access Criteria: Scientific researchers interested in obtaining the protocol, statistical analysis plan, informed consent form, or clinical study report for educational purposes or to participate in the trial can request these materials by contacting the principal investigator or study coordinator.

REFERENCES:
- [Background] Ryan JF, Motz KM, Rooper LM, Mydlarz WK, Quon H, Gourin CG, Tan M, Eisele DW, Fakhry C. The Impact of a Stepwise Approach to Primary Tumor Detection in Squamous Cell Carcinoma of the Neck With Unknown Primary. Laryngoscope. 2019 Jul;129(7):1610-1616. doi: 10.1002/lary.27625. Epub 2018 Nov 22. PMID 30565698
- [Background] Chaturvedi AK, Anderson WF, Lortet-Tieulent J, Curado MP, Ferlay J, Franceschi S, Rosenberg PS, Bray F, Gillison ML. Worldwide trends in incidence rates for oral cavity and oropharyngeal cancers. J Clin Oncol. 2013 Dec 20;31(36):4550-9. doi: 10.1200/JCO.2013.50.3870. Epub 2013 Nov 18. PMID 24248688
- [Background] Ren J, Yang W, Su J, Ren X, Fazelzad R, Albert T, Habbous S, Goldstein DP, de Almeida JR, Hansen A, Jang R, Bratman SV, Hope A, Chen R, Wang J, Xu Y, Cheng D, Zhao Y, Xu W, Liu G. Human papillomavirus and p16 immunostaining, prevalence and prognosis of squamous carcinoma of unknown primary in the head and neck region. Int J Cancer. 2019 Sep 15;145(6):1465-1474. doi: 10.1002/ijc.32164. Epub 2019 Feb 19. PMID 30698281
- [Background] Chen B, Zhang H, Liu D, Wang X, Ji B, Gao S. Diagnostic performance of 18F-FDG PET/CT for the detection of occult primary tumors in squamous cell carcinoma of unknown primary in the head and neck: a single-center retrospective study. Nucl Med Commun. 2021 May 1;42(5):523-527. doi: 10.1097/MNM.0000000000001365. PMID 33481505
- [Background] Farooq S, Khandavilli S, Dretzke J, Moore D, Nankivell PC, Sharma N, Almeida JR, Winter SC, Simon C, Paleri V, De M, Siddiq S, Holsinger C, Ferris RL, Mehanna H. Transoral tongue base mucosectomy for the identification of the primary site in the work-up of cancers of unknown origin: Systematic review and meta-analysis. Oral Oncol. 2019 Apr;91:97-106. doi: 10.1016/j.oraloncology.2019.02.018. Epub 2019 Mar 6. PMID 30926070
- [Background] Maghami E, Ismaila N, Alvarez A, Chernock R, Duvvuri U, Geiger J, Gross N, Haughey B, Paul D, Rodriguez C, Sher D, Stambuk HE, Waldron J, Witek M, Caudell J. Diagnosis and Management of Squamous Cell Carcinoma of Unknown Primary in the Head and Neck: ASCO Guideline. J Clin Oncol. 2020 Aug 1;38(22):2570-2596. doi: 10.1200/JCO.20.00275. Epub 2020 Apr 23. PMID 32324430
- [Background] Ferris RL, Flamand Y, Weinstein GS, Li S, Quon H, Mehra R, Garcia JJ, Chung CH, Gillison ML, Duvvuri U, O'Malley BW Jr, Ozer E, Thomas GR, Koch WM, Gross ND, Bell RB, Saba NF, Lango M, Mendez E, Burtness B. Phase II Randomized Trial of Transoral Surgery and Low-Dose Intensity Modulated Radiation Therapy in Resectable p16+ Locally Advanced Oropharynx Cancer: An ECOG-ACRIN Cancer Research Group Trial (E3311). J Clin Oncol. 2022 Jan 10;40(2):138-149. doi: 10.1200/JCO.21.01752. Epub 2021 Oct 26. PMID 34699271
- [Background] Chen AM. De-Escalation Treatment for Human Papillomavirus-Related Oropharyngeal Cancer: Questions for Practical Consideration. Oncology (Williston Park). 2023 Jul 21;37(7):281-287. doi: 10.46883/2023.25921000. PMID 37499250
- [Background] Sivars L, Nasman A, Tertipis N, Vlastos A, Ramqvist T, Dalianis T, Munck-Wikland E, Nordemar S. Human papillomavirus and p53 expression in cancer of unknown primary in the head and neck region in relation to clinical outcome. Cancer Med. 2014 Apr;3(2):376-84. doi: 10.1002/cam4.199. Epub 2014 Feb 10. PMID 24510528
- [Background] Mackenzie K, Watson M, Jankowska P, Bhide S, Simo R. Investigation and management of the unknown primary with metastatic neck disease: United Kingdom National Multidisciplinary Guidelines. J Laryngol Otol. 2016 May;130(S2):S170-S175. doi: 10.1017/S0022215116000591. PMID 27841129
- [Background] Network NCC. 2023. NCCN clinical practice guidelines in oncology: head and neck cancers. Fort Washington, PA, nd.
- [Background] Axelsson L, Nyman J, Haugen-Cange H, Bove M, Johansson L, De Lara S, Kovacs A, Hammerlid E. Prognostic factors for head and neck cancer of unknown primary including the impact of human papilloma virus infection. J Otolaryngol Head Neck Surg. 2017 Jun 10;46(1):45. doi: 10.1186/s40463-017-0223-1. PMID 28601094
- [Background] Wichmann G, Willner M, Kuhnt T, Kluge R, Gradistanac T, Wald T, Fest S, Lordick F, Dietz A, Wiegand S, Zebralla V. Standardized Diagnostics Including PET-CT Imaging, Bilateral Tonsillectomy and Neck Dissection Followed by Risk-Adapted Post-Operative Treatment Favoring Radio-Chemotherapy Improve Survival of Neck Squamous Cell Carcinoma of Unknown Primary Patients. Front Oncol. 2021 May 7;11:682088. doi: 10.3389/fonc.2021.682088. eCollection 2021. PMID 34026656
- [Background] Zhou MJ, van Zante A, Lazar AA, Groppo ER, Garsa AA, Ryan WR, El-Sayed IH, Eisele DW, Yom SS. Squamous cell carcinoma of unknown primary of the head and neck: Favorable prognostic factors comparable to those in oropharyngeal cancer. Head Neck. 2018 May;40(5):904-916. doi: 10.1002/hed.25028. Epub 2017 Dec 6. PMID 29210145
- [Background] Takhar A, Wilkie MD, Srinivasan D, King E. Head and Neck Squamous Cell Carcinoma of Unknown Primary-Who Can Be Offered Surgery as the Sole Treatment Modality? A Systematic Review. Clin Otolaryngol. 2025 May;50(3):399-414. doi: 10.1111/coa.14279. Epub 2025 Jan 12. PMID 39800989
- [Background] Strojan P, Kokalj M, Zadnik V, Anicin A, Plavc G, Didanovic V, Sifrer R, Lanisnik B. Squamous cell carcinoma of unknown primary tumor metastatic to neck nodes: role of elective irradiation. Eur Arch Otorhinolaryngol. 2016 Dec;273(12):4561-4569. doi: 10.1007/s00405-016-4172-5. Epub 2016 Jun 30. PMID 27363402
- [Background] Poon WY, Thomson M, McLoone P, Wilson C, Crosbie R, Schipani S, Grose D, James A, Lamb C, Rizwanullah M, Campbell F, Easton F, Paterson C. Comparative cohort study of volumetric modulated arc therapy for squamous cell cancer of unknown primary in the head and neck-Involved neck only versus mucosal irradiation. Clin Otolaryngol. 2020 Nov;45(6):847-852. doi: 10.1111/coa.13593. Epub 2020 Sep 17. PMID 32501648
- [Background] Grewal AS, Rajasekaran K, Cannady SB, Chalian AA, Ghiam AF, Lin A, LiVolsi V, Lukens JN, Mitra N, Montone KT, Newman JG, O'Malley BW Jr,, Rassekh CH, Weinstein GS, Swisher-McClure S. Pharyngeal-sparing radiation for head and neck carcinoma of unknown primary following TORS assisted work-up. Laryngoscope. 2020 Mar;130(3):691-697. doi: 10.1002/lary.28200. Epub 2019 Aug 14. PMID 31411747
- [Background] Patel MR, Ottenstein L, Ryan M, Farrell A, Studer M, Baddour HM, Magliocca K, Griffith C, Stokes W, Switchenko J, Aiken A, El-Deiry M, Solares CA, Steuer C, Saba N, Beitler J. TORS elective lingual tonsillectomy has less acute morbidity than therapeutic base of tongue TORS. Oral Oncol. 2021 Jun;117:105294. doi: 10.1016/j.oraloncology.2021.105294. Epub 2021 Apr 17. PMID 33878679
- [Background] Swiecicki PL, Bellile E, Dragovic AF, McHugh J, Udager A, Mierzwa ML, Shah J, Heft-Neal M, Rosko A, Malloy KM, Casper K, Chinn SB, Shuman AG, Stucken C, Chepeha DB, Wolf GT, Bradford CR, Eisbruch A, Prince ME, Worden FP, Spector ME. Upfront Neck Dissection for Treatment Selection and Improvement in Quality of Life as a Novel Treatment Paradigm for Deintensification in HPV+ OPSCC. Clin Cancer Res. 2024 Jun 3;30(11):2393-2401. doi: 10.1158/1078-0432.CCR-23-3247. PMID 38517480
- [Background] Lauer MS, D'Agostino RB Sr. The randomized registry trial--the next disruptive technology in clinical research? N Engl J Med. 2013 Oct 24;369(17):1579-81. doi: 10.1056/NEJMp1310102. Epub 2013 Aug 31. No abstract available. PMID 23991657